CLINICAL TRIAL: NCT00419120
Title: An Open-Label Multicenter Study of Augmentation Cystoplasty Using an Autologous Neo-Bladder Construct in Subjects With Spina Bifida
Brief Title: Augmentation Cystoplasty Using an Autologous Neo-Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 36 months follow up without change to profile. No further studies planned.
Sponsor: Tengion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNG-CL003
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neo-bladder construction (Experimental): Surgical implantation of autologous neo-bladder construct
  Interventions: Biological: Autologous neo bladder construct

INTERVENTIONS:
Biological: Autologous neo bladder construct — augmentation cystoplasty with autologous neo-bladder construct

SUMMARY:
Subjects with neurogenic bladder secondary to spina bifida refractory to medical treatment will be enrolled. The hypothesis is that augmentation cystoplasty using an autologous neo-bladder construct will significantly increase bladder compliance.

DETAILED DESCRIPTION:
Subjects with neurogenic bladder secondary to spina bifida (myelodysplasia) that is refractory to medical treatment and require augmentation cystoplasty will be enrolled. The hypothesis is that augmentation cystoplasty using an autologous neo-bladder construct will significantly increase bladder compliance.

ELIGIBILITY:
Inclusion Criteria:

* subjects with neurogenic bladders secondary to myleodysplasia

Exclusion Criteria:

* prior augment procedures
* recent urologic surgery
* requires concomitant urologic intervention

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Sheth, MD, Study Director — Tengion, Inc.
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were recruited between Dec 2006 and July 2007. Patients were recruited from 4 academic centers across the US. One patient withdrew from the study prior to implantation of the Neo-bladder construct and is included in the safety analysis, but not in the efficacy analysis (all implanted population).
Pre-assignment Details: This was an open label single arm study.
Groups:
- Implanted Patients: Patients implanted with Tengion Neo-Bladder Augment
Period: Primary Study Period
Arm/Group | Implanted Patients
Started | 10
Completed | 10
Not Completed | 0
Period: Long Term Follow up Period
Arm/Group | Implanted Patients
Started | 10 (10 patients are being followed in long term follow up.)
Completed | 0
Not Completed | 10
Not completed — study ongoing | 10

BASELINE CHARACTERISTICS:
Arm/Group | Implanted Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders as Assessed by Compliance
Description: Efficacy of the autologous neo-bladder construct as assessed by a responder analysis (comparing each patient's baseline with 12 month data). Improvement in compliance (i.e. improved bladder pressure/volume relationship) was measured by urodynamics at predetermined bladder pressure points. This was coupled with an assessment of clinical benefit and used to determine responders versus non-responders
Time Frame: 12 months
Population: The analysis population of the primary outcome measure is the all implanted population (Intent to Treat - ITT). There was no imputation of analysis measures.
Measure: Number; unit: participants
Arm/Group | Implanted Patients
Number analyzed (Participants) | 10
participants | 6

2. Secondary Outcome: Overall Safety Profile - Number of Participants Experiencing an Adverse Event
Description: clinical evaluation of adverse events, laboratory parameters and urinary imaging to assess any safety issues emerging from this technology and to allow a comparison of a safety profile with standard of care enterocystoplasty. Please refer to the Adverse Event section for detailed information.
Time Frame: periodically within first 12 months as well as during long term follow up out to 5 years
Measure: Number; unit: participants
Arm/Group | Implanted Patients
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Description: Adverse events are reported for 11 subjects who were enrolled in the study. One patient withdrew prior to implantation with the neo-bladder construct and is included in the safety population but not in the all implanted population used for efficacy analysis.
Groups:
- Safety Population: All patients undergoing screeing and meeting inclusion/exclusion criteria
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=11)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Ventriculoperitoneal Shunt Malfunction (Injury, poisoning and procedural complications) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Complication of Device Insertion (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Urine Leak (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Implant Site Inflammation (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 10 (37)
Nasopharyngitis (Infections and infestations) | 3 (4)
Clostridial Infection (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Enterococcal Infection (Infections and infestations) | 1 (1)
Molluscum Contagiosum (Infections and infestations) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1)
Hemoglobin Decreased (Investigations) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (4)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator is free to individually communicate, orally present or publish in scientific journals or other scholarly media the study information at the conclusion of the study without the prior approval of the sponsor provided that 1)the results of the study in its entirely have been publically disclosed by or with the consent of the sponsor 2)18 months after the conclusion of the study at all sites whichever is first to occur.